CLINICAL TRIAL: NCT05775315
Title: Additional Effects of Visual Feedback Along With Action Observation Therapy on Balance, Mobility and Cognition in Cerebral Palsy
Brief Title: Additional Effect of Visual Feedback Along With AOT on Balance,Mobility and Cognition in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01363 Ayesha Tabassum
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy
Keywords: action observation therapy; cerebral palsy; visual feedback
MeSH Terms: conditions — Cerebral Palsy | interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy (Experimental): exercises of AO protocol
  Interventions: Other: Action Observation Therapy
- Visual feedback and Action Observation Therapy (Active Comparator): Excercises of AO protocol infront of a mirror
  Interventions: Other: Action Observation Therapy along with visual feedback

INTERVENTIONS:
Other: Action Observation Therapy — Exercises of AO protocol MOVEMENT TOTAL VIDEO TIME PATIENT TIME Upright the pelvis 1 minute 5 minutes Move weight forward 1 minute 5 minutes Move weight to the left and right 1 minute 5 minutes Rotate right and left 1 minute 5 minutes Upright the pelvis in sitting position 1 minute 5 minutes Move weight forward from a sitting position 1 minute 5 minutes Stand up from a sitting position 1 minute 5 minutes Move weight right and left 1 minute 5 minutes Forward weight shift with right foot and left foot 1 minute 5 minutes Walking sideways to left 1 minute 5 minutes Walking sideways to right 1 minute 5 minutes
  Rest time between watching and performing each video will be 1 minute. the exercises will be done 3 times a week.
  Arms: Action Observation Therapy
Other: Action Observation Therapy along with visual feedback — Exercises of AO protocol in front of a mirror MOVEMENT TOTAL VIDEO TIME PATIENT TIME Upright the pelvis 1 minute 5 minutes Move weight forward 1 minute 5 minutes Move weight to the left and right 1 minute 5 minutes Rotate right and left 1 minute 5 minutes Upright the pelvis in sitting position 1 minute 5 minutes Move weight forward from a sitting position 1 minute 5 minutes Stand up from a sitting position 1 minute 5 minutes Move weight right and left 1 minute 5 minutes Forward weight shift with right foot and left foot 1 minute 5 minutes Walking sideways to left 1 minute 5 minutes Walking sideways to right 1 minute 5 minutes
  Rest time between watching and performing each video will be 1 minute. the exercises will be done 3 times a week.
  Arms: Visual feedback and Action Observation Therapy

SUMMARY:
the study aims to find the effectiveness of visual feedback along with action observation therapy in cerebral palsy. the effect of AOT on mobility, cognition and balance of the targeted population will be the intrest of the researcher

ELIGIBILITY:
Inclusion Criteria:

* Without visual impairment and visual field defects
* Mini-Mental state examination for Children (MMC) score >25
* GMFCS (gross motor function classification system) I-III
* Children with Modified Ashworth Scale (MAS) less than 2

Exclusion Criteria:

* Unable to walk
* Children with severe co-morbidities

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification Scale (GMFCS) | 12 weeks
  Gross Motor Function measure (GMFM) is the valid and standard observational instrument to measure change in gross motor function in CP children. The tool consists of 66 items with 5 dimensions. These dimensions are the major motor functions i.e. supine/rolling, sitting, crawling/kneeling, standing and walking/running/jumping. Each task is rated according to the scoring guidelines i.e. higher score indicated better gross motor function. Each GMFM item is graded on 4-point scale i.e. 0 for unable to initiate the task, 1 for able to initiate the task, 2 for able to perform the task partially and 3 for able to perform the task completely. At the end these score summed up into total score. The component B,C,D and E of GMFCS will be used in this study respectively.
Pediatric Balance Scale (PBS) | 12 weeks
  PBS is a modified form of Berg Balance Scale (BSS) which was developed for balance measurement in CP child. It can be performed without specialized equipment and is easy to administrate. It includes 14 items with 5-level grading to assess the functional activities that child must safely and independently form at home, community, activities including sitting balance, sit to stand/stand to sit, transfer, stepping, reaching forward, reaching to floor, turning and stepping on and off at elevated surface. Each activity is rated according to scale from 0 to 4 i.e. 0 for unable to perform and 4 for able to perform without difficulty.
Timed 10-meter walk test | 12 weeks
  The test can be used to measure the gait ability and speed. The acceleration area 2.5m and deceleration area 2.5m can be marked on the ground as start and end point for the test. Participants are asked to walk for 15 minutes on comfortable flat floor at a comfortable speed and then the walking speed is recorded through stopwatch over 10 m between these points. The mean value of the three trials was used and expressed as m/s(14).
Mini Mental State Exam | 12 weeks
  It is a cognitive screening task and scoring system for 3 to 14 years old child (25). It is presented by 11 questions involving five basic cognitive abilities i.e. attention-concentration, orientation, registration, recall and language and constructive ability. The possible score range is from 0 to 37, from which 17 or lower score indicating as moderate to severe cognitive impairment of children.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Bashir, Principal Investigator — Riphah International University
Locations (1):
- Center for Profound Education Trust, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arliani GG, Astur DC, Yamada RK, Yamada AF, da Rocha Correa Fernandes A, Ejnisman B, de Castro Pochini A, Cohen M. Professional football can be considered a healthy sport? Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3907-3911. doi: 10.1007/s00167-015-3636-2. Epub 2015 May 17. PMID 25982623
- [Background] Bell DR, Guskiewicz KM, Clark MA, Padua DA. Systematic review of the balance error scoring system. Sports Health. 2011 May;3(3):287-95. doi: 10.1177/1941738111403122. PMID 23016020
- [Background] Hoffer ME, Gottshall KR, Moore R, Balough BJ, Wester D. Characterizing and treating dizziness after mild head trauma. Otol Neurotol. 2004 Mar;25(2):135-8. doi: 10.1097/00129492-200403000-00009. PMID 15021772
- [Background] Gurr B, Moffat N. Psychological consequences of vertigo and the effectiveness of vestibular rehabilitation for brain injury patients. Brain Inj. 2001 May;15(5):387-400. doi: 10.1080/02699050010005904. PMID 11350653
- [Background] Murray DA, Meldrum D, Lennon O. Can vestibular rehabilitation exercises help patients with concussion? A systematic review of efficacy, prescription and progression patterns. Br J Sports Med. 2017 Mar;51(5):442-451. doi: 10.1136/bjsports-2016-096081. Epub 2016 Sep 21. PMID 27655831
- [Background] Balatsouras DG, Koukoutsis G, Aspris A, Fassolis A, Moukos A, Economou NC, Katotomichelakis M. Benign Paroxysmal Positional Vertigo Secondary to Mild Head Trauma. Ann Otol Rhinol Laryngol. 2017 Jan;126(1):54-60. doi: 10.1177/0003489416674961. Epub 2016 Oct 25. PMID 27780909
- [Background] McCrea M, Guskiewicz KM, Marshall SW, Barr W, Randolph C, Cantu RC, Onate JA, Yang J, Kelly JP. Acute effects and recovery time following concussion in collegiate football players: the NCAA Concussion Study. JAMA. 2003 Nov 19;290(19):2556-63. doi: 10.1001/jama.290.19.2556. PMID 14625332
- [Background] Alsalaheen BA, Mucha A, Morris LO, Whitney SL, Furman JM, Camiolo-Reddy CE, Collins MW, Lovell MR, Sparto PJ. Vestibular rehabilitation for dizziness and balance disorders after concussion. J Neurol Phys Ther. 2010 Jun;34(2):87-93. doi: 10.1097/NPT.0b013e3181dde568. PMID 20588094
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] O'Connor KL, Rowson S, Duma SM, Broglio SP. Head-Impact-Measurement Devices: A Systematic Review. J Athl Train. 2017 Mar;52(3):206-227. doi: 10.4085/1062-6050.52.2.05. PMID 28387553
- [Background] Clark MD, Asken BM, Marshall SW, Guskiewicz KM. Descriptive Characteristics of Concussions in National Football League Games, 2010-2011 to 2013-2014. Am J Sports Med. 2017 Mar;45(4):929-936. doi: 10.1177/0363546516677793. Epub 2017 Jan 5. PMID 28056179
- [Background] Broglio SP, Collins MW, Williams RM, Mucha A, Kontos AP. Current and emerging rehabilitation for concussion: a review of the evidence. Clin Sports Med. 2015 Apr;34(2):213-31. doi: 10.1016/j.csm.2014.12.005. Epub 2015 Jan 24. PMID 25818710
- [Background] Gasquoine PG. Historical perspectives on evolving operational definitions of concussive brain injury: From railway spine to sport-related concussion. Clin Neuropsychol. 2020 Feb;34(2):278-295. doi: 10.1080/13854046.2019.1621383. Epub 2019 May 31. PMID 31146639